CLINICAL TRIAL: NCT01975779
Title: Interventional, Randomised, Double-blind, Placebocontrolled, Single- and Multiple-ascending-dose Study Investigating the Safety, Tolerability, and Pharmacokinetic Properties of Lu AE58054 in Healthy Japanese and Caucasian Subjects
Brief Title: Study Investigating the Safety, Tolerability, and Pharmacokinetic Properties of Lu AE58054 in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14917A; 2012-005648-10 (EudraCT Number)
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A1: Lu AE58054 or placebo (Experimental)
  Interventions: Drug: Cohort A1: Lu AE58054 or placebo
- Cohort A2: Lu AE58054 or placebo (Experimental)
  Interventions: Drug: Cohort A2: Lu AE58054 or placebo
- Cohort B1: Lu AE58054 (Experimental)
  Interventions: Drug: Cohort B1: Lu AE58054

INTERVENTIONS:
Drug: Cohort A1: Lu AE58054 or placebo — One single oral dose 60 mg (one 60 mg tablet) followed by 60 mg once daily for 7 days, or matching placebo.
  Arms: Cohort A1: Lu AE58054 or placebo
Drug: Cohort A2: Lu AE58054 or placebo — One single oral dose 120 mg (two 60 mg tablets) followed by 120 mg once daily for 7 days, or matching placebo.
  Arms: Cohort A2: Lu AE58054 or placebo
Drug: Cohort B1: Lu AE58054 — Two single oral doses 60 mg with >=7 days washout.
  Arms: Cohort B1: Lu AE58054

SUMMARY:
To evaluate the safety and tolerability of single- and multiple doses of Lu AE58054 in healthy young Japanese men in comparison with Caucasian men.

DETAILED DESCRIPTION:
The study will be conducted in two parts.

Part A consists of two cohorts (named cohort A1 and A2), which are randomised, double-blind, parallel-group, placebo-controlled, single- and multiple dose regimens investigating the safety, tolerability, and pharmacokinetics of Lu AE58054 in healthy young men.

Part B consists of one cohort, B1, which is a randomised, open-label, two-way cross-over, single dose investigation of the effect of food on the pharmacokinetics of Lu AE58054 in healthy young Japanese men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese (Japanese passport, four Japanese grandparents, and lives outside Japan for less than 5 years) or Caucasian men aged 20 to 45 years with a BMI between 18 and 25 kg/m2 (extremes included).

Exclusion Criteria:

* The subject is, in the opinion of the investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.

Other inclusion and exclusion criteria may apply.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number and frequency of adverse events | Up to Day 13
  Standard clinical safety assessments
Number of subjects with adverse events | Up to Day 13
  Adverse event monitoring

SECONDARY OUTCOMES:
Area under the Lu AE58054 plasma concentration-time curve in a dosing interval (AUC0-tau) | Day 9
Area under the Lu AE58054 plasma concentration-time curve from zero to infinity (AUC0-inf) | Day 1
Maximum observed concentration (Cmax) and time of observation (tmax) | Day 1 and Day 9
Oral clearance (CL/F), apparent volume of distribution (Vz/F), and elimination halflife (t½) | Day 1 and Day 9
Accumulation index following multiple dosing of Lu AE58054 (AI) | Day 9
Risk of Suicidality | Up to Day 13
  Columbia Suicide Severity Rating Scale (C-SSRS) categorisation based on Columbian Classification Algorithm for Suicide Assessment (C-CASA) definitions for Part A

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- GB001, London, United Kingdom